CLINICAL TRIAL: NCT06201299
Title: Comparison of the Effectiveness of Chair-based and Standard Exercise Programs in People With COPD
Brief Title: Chair-based and Standard Exercise Programs in People With COPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, esra pehlivan, Assoc. Prof. Dr., Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COPD_Chair exercises
Record Dates: First submitted 2023-12-30; First posted 2024-01-11 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: COPD; Pulmonary Rehabilitation; Exercise
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chair-based Exercise Group (Experimental): Exercises will be performed with chair support.
  Interventions: Other: Chair-based Exercise Program
- Standard Exercise Group (Experimental): Exercises will be performed using theraband.
  Interventions: Other: Standard Exercise Program

INTERVENTIONS:
Other: Standard Exercise Program — The program content consists of breathing exercises, upper and lower extremity strengthening with theraband and self-walking. Chest, abdominal and lateral basal breathing exercises will be performed 10 times each. Resistance exercises will be performed as strengthening exercises for the major muscle groups of the upper and lower extremities using medium-hard theraband. Patients will be asked to walk 30 minutes a day on flat ground at 60% workload, for periods calculated according to the 6-minute walk test results (land-based walking).
  Arms: Standard Exercise Group
Other: Chair-based Exercise Program — The program content consists of breathing exercises and chair-supported exercises. Chest, abdominal and lateral basal breathing exercises will be performed 10 times each. Chair exercises are given in the exercise brochure. Exercises are performed with a chair support or sitting on a chair. In addition, patients will be asked to walk 30 minutes a day on flat ground at 60% workload, for periods calculated according to the 6-minute walk test results (land-based walking).
  Arms: Chair-based Exercise Group

SUMMARY:
Patients who are diagnosed with COPD by a pulmonology specialist and referred to pulmonary rehabilitation will be included in the study. Cases that meet the inclusion criteria will be randomized and divided into two groups, standard exercise program group (SGr) and chair-based exercise. program group will be called (ChGr). While standard exercises will be given to SGr, chair-based exercises will be applied to ChGr. All evaluation and initial training sessions of the cases will be held in the hospital. Apart from this, they will be asked to do their exercises at home with the exercise videos that will be sent to them. In order to ensure that home exercises are performed completely and correctly, 2 sessions of online simultaneous exercise training will be provided with a physiotherapist via videoconference on a smartphone, and exercise follow-ups will be carried out by calling once a week. The program duration is 8 weeks, 5 days a week.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-75 years
* Having a diagnosis of COPD diagnosed according to clinical diagnostic criteria according to the American Thoracic and European Respiratory Societies (ATS-ERS).
* Presence of dyspnea on exertion
* Stable clinical status at inclusion without infection or exacerbation in the previous 4 weeks *Having smart phone usage skills

Exclusion Criteria:

* Patients with severe comorbid diseases, unstable coronary artery disease, collagen vascular diseases and requiring high-flow oxygen therapy (˃ 3-4 L\min).
* A history of exertional syncope or the presence of any comorbidities (such as severe orthopedic or neurological deficits or unstable heart disease) that preclude exercise training.
* Having participated in a pulmonary rehabilitation program within the last 12 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-01-20 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Exercise capacity assesment | Change from baseline at 2 months
  The 6-minute walking test will conduct in a 30-meter corridor in line with American Thoracic Society (ATS) guidelines. Participants will ask to walk as far as they can. Prior to and following the test, oxygen saturation, heart rate and Borg fatigue rating will measure, and the walking distance will record.

SECONDARY OUTCOMES:
Dyspnea evaluation | Change from baseline at 2 months
  Modified Medical Council Dyspnea score will rate the sensation of dyspnea as the person perceives it.The severity of dyspnea is rated on a scale of 0 to 4."0 point" means no dyspnea perception and "4point" means severe dyspnea perception.
Respiratory muscle strength measurement | Change from baseline at 2 months
  The mouth pressure measurement (maximum inspiratory and expiratory pressure) will perform with the Pony Fx spirometry device. Patient will place a rubber mouthpiece with flanges, on the device, exhale/inhale slowly and completely, and then will try to breath in as hard as possible. The patient will allow to rest for about a minute and the maneuver will repeat. The aim is that the variability between measurements is less than 10 cm H2O. The maximum value will obtain.
Peripheral muscle strength measurement | Change from baseline at 2 months
  Strength measurements of major peripheral muscle groups will be made with a digital myometer.
Evaluation of quality of life | Change from baseline at 2 months
  Saint George Respiratory Questionaire (SGRQ) score: The SGRQ ranges from 0 (no impairment of quality of life) to 100 (highest impairment of quality of life).
Evaluation of fatigue | Change from baseline at 2 months
  The fatigue severity scale: A 9-item questionnaire with questions related to how fatigue interferes with certain activities and rates its severity.
  The items are scored on a 7 point scale with 1 = strongly disagree and 7= strongly agree The minimum score = 9 and maximum score possible = 63. Higher the score = greater fatigue severity Another way of scoring: mean of all the scores with minimum score being 1 and maximum score being 7 Self-report scale
Psychological status assessment | Change from baseline at 2 months
  Hospital Anxiety Depression scale:The levels of anxiety and depression will asses by Hospital Anxiety Depression Scale (HADS) .The HADS is a self-report rating scale of 14 items on a 4-point Likert scale (range 0-3). It is designed to measure anxiety and depression (7 items for each subscale). The total score is the sum of the 14 items, and for each subscale the score is the sum of the respective seven items (ranging from 0-21).Several studies suggest a cut-off score of ≥8 to be optimal for best sensitivity and specificity. The HADS has sensitivity and specificity of about 80%, and a predictive validity for identification of about 70%.
Physical activity level assesment | Change from baseline at 2 months
  The International Physical Activity Questionnaire (IPAQ) was developed as an instrument for cross-national monitoring of physical activity and inactivity. This measure assesses the types of intensity of physical activity and sitting time that people do as part of daily lives are considered to estimate total physical activity in MET-min/week and time spent sitting.
Pulmonary function tests (PFTs) | Change from baseline at 2 months
  PFTs will perform by using the Pony Fx spirometry device, and according to the American Thoracic Society (ATS) guidelines

CONTACTS AND LOCATIONS:
Locations (1):
- Yedikule Chest Disease Hospital, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided